CLINICAL TRIAL: NCT04740645
Title: Post-authorisation Safety Study of NOCDURNA for the Symptomatic Treatment of Nocturia Due to Idiopathic Nocturnal Polyuria: A Multi-country Cohort Study Using Secondary Data
Brief Title: NOCDURNA PASS Study Using Registries in Denmark, Germany and Sweden
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000248
Record Dates: First submitted 2021-01-29; First posted 2021-02-05 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Adverse Drug Event
Keywords: Nocturia; NOCDURNA; Post-authorisation Safety Study
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Nocturia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NOCDURNA cohort
  Interventions: Other: NOCDURNA Cohort
- Lower urinary tract symptoms (LUTS) Cohort
  Interventions: Other: LUTS Cohort

INTERVENTIONS:
Other: NOCDURNA Cohort — Non intervention
  Groups: NOCDURNA cohort
Other: LUTS Cohort — Non intervention
  Groups: Lower urinary tract symptoms (LUTS) Cohort

SUMMARY:
A study using medical records to evaluate safety issues for the NOCDURNA drug using national register data from Denmark and Sweden, and a health care register covering parts of Germany.

ELIGIBILITY:
Inclusion Criteria:

* Usage of NOCDURNA recorded as dispensations in adults or usage of drugs for LUTS.

Exclusion Criteria:

* Multiple dispensations of NOCDURNA on the same day or treatment with vasopressin 6 months before study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with usage of NOCDURNA identified as dispensations/prescriptions or dispensations/prescription of drugs for LUTS
Sampling Method: Non-Probability Sample
Enrollment: 1099551 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence rate of symptomatic hyponatraemia | Through study completion, typically 2 months
  Symptomatic hyponatraemia was defined as a primary or secondary diagnosis of hyponatraemia.

SECONDARY OUTCOMES:
Incidence rate of hyponatraemia requiring hospital intensive care | Through study completion, typically 2 months
  Hyponatraemia requiring hospital intensive care was defined as a primary or secondary diagnosis of hyponatraemia recorded in an intensive care unit.
Incidence and severity of clinically significant hyponatraemia | Through study completion, typically 2 months
  Clinically significant hyponatraemia was defined as a serum sodium concentration of <130 mmol/L. Severity of hyponatraemia was categorized as mild hyponatraemia (serum sodium concentration: 130 to <135 mmol/L), moderate hyponatraemia (serum sodium concentration: >125 to <130 mmol/L) and severe hyponatraemia (serum sodium concentration: less than equal to [≤]125 mmol/L).
Rate of all-cause mortality | Through study completion, typically 2 months
  All-cause mortality was defined as death from any cause.
Incidence rate of major adverse cardiovascular events (MACE) | Through study completion, typically 2 months
  Major adverse cardiovascular events were defined as a record of myocardial infarction and stroke. Fatal and non-fatal events will be considered separately.
Incidence rate of major venous thromboembolic events (VTEs) | Through study completion, typically 2 months
  Venous thromboembolic events were defined as a record of a deep vein thrombosis, pulmonary embolism or portal vein thrombosis. Fatal and non-fatal events will be considered separately.
Incidence rate acute exacerbation of congestive heart failure | Through study completion, typically 2 months
  Acute exacerbation of congestive heart failure was defined as primary diagnosis of acute or acute-on-chronic heart failure from hospital inpatient care or the acute and emergency ward, or death from heart failure as the underlying or contributory cause.
Incidence of serious adverse events of MACE and VTE in Sweden | Through study completion, typically 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (3):
- Danish Health Care Registry, Copenhagen, Denmark
- German Health Care Register, Bremen, Germany
- Socialstryrelsen, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Johansson G, Reinold J, Shapero NL, Rosell TL, Jorgensen LA, Koenen N, Frosig C, Falkenberg M, Holdrup L, Juul K. Real-life safety assessment of orally disintegrating desmopressin tablet: Incidence of diagnosed hyponatraemia and other events across three European countries. Glob Epidemiol. 2025 Oct 31;10:100228. doi: 10.1016/j.gloepi.2025.100228. eCollection 2025 Dec. PMID 41281576
- See also: DOI: 10.1016/j.gloepi.2025.100228 — https://doi.org/10.1016/j.gloepi.2025.100228